CLINICAL TRIAL: NCT06428929
Title: The Effect of Using Musical and Lighted Baby Crib Mobile on Newborns' Pain and Stress During Blood Draw: Randomized Controlled Trial
Brief Title: The Effect of Using Musical and Lighted Baby Crib Mobile on Newborns' Pain and Stress During Blood Draw
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Eysan Hanzade Umac, Research Assistant, Koç University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EysanUmac
Record Dates: First submitted 2024-05-15; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Newborns were randomly assigned groups as the musical and lighted baby crib mobile (intervention) group (40 newborns) and the control group (40 newborns) by the computer program (www.randomizer.org). Newborns of parents who did not meet the study criteria and did not agree to participate in the random selection were not included in the study. Parents and researchers could not be blinded. Newborns were included in the study by evaluating their compliance with the inclusion criteria according to the order of admission to the hospital. 10 children in the control group (5 parents did not volunteer and 5 newborns were crying) and 10 children in the intervention group (7 newborns received paracetamol and 3 newborns were crying) were excluded from the study. For this reason, the research was completed with 60 newborns.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Infants in the control group received standard care, with no pharmacological or non-pharmacological methods used to reduce pain, except for allowing the parents to be present. Parents and nurses observed the infant's behavior during and immediately after the procedure to assess pain and stress. After the procedure, they were asked to mark the maximum pain and stress experienced by the baby on the "ALPS-Neo pain and stress rating scale." This assessment was done immediately after the needle was removed and a tampon was placed to stop the bleeding, approximately one minute after the procedure.
- Intervention (Experimental): Before the procedure, the researcher informed the parents of the newborns in the musical and lighted baby crib mobile group about the study procedure and purpose. The mobile was fixed 60 cm above the newborn's eye level to prevent contamination and trauma. After obtaining written consent, the researcher collected data using the 'Newborn Information Form' through face-to-face interviews. Once the form was completed, the mobile was activated. One minute later, the nurse performed the blood draw. Parents and nurses observed the infant's behavior during and immediately after the procedure to assess pain and stress. They were then asked to mark the maximum pain and stress experienced by the baby on the ALPS-Neo pain and stress rating scale.
  Interventions: Other: The musical and lighted baby crib mobile:

INTERVENTIONS:
Other: The musical and lighted baby crib mobile: — The musical and lighted baby crib mobile: It measures 43.5x33x9.5 cm and is made of plastic. It is recommended for use in infants 0-12 months. It has music that makes it easier for babies to fall asleep by reducing stress. This baby mobile has a projection and music function. In addition, the mobile has a 360° flexible swivel bracket that can be adjusted as desired. The surface of the apparatus of the mobile, which is designed to be environmentally and baby friendly, is smooth. There are four rattles on the mobile
  Arms: Intervention

SUMMARY:
It is widely recognized that the use of non-pharmacological methods in neonatal pain management is low both globally and in our country. Nurses play a crucial role in managing pain through various techniques and in preventing its negative effects on newborns. Toys with sounds, lights, and different features have been found to effectively capture infants' attention. Consequently, it is anticipated that baby crib mobiles, which combine these attention-grabbing features, could serve as effective distractions during needle interventions, potentially reducing pain and stress. However, there is a lack of research on this specific application.

DETAILED DESCRIPTION:
Newborns often undergo needle procedures shortly after birth, such as vitamin K injections, hepatitis B vaccinations, screenings, and routine immunizations. Depending on the baby's condition, these procedures may need to be repeated, and additional blood samples might be required. These painful procedures can cause significant stress for the newborn and may lead to neurocognitive, physiological, metabolic, and behavioral issues. Pain experienced during these procedures can negatively impact the newborn's future reactions to pain. Therefore, inadequate pain management can result in both immediate and long-term adverse effects.

Organizations such as the International Neuropsychiatric Pain Group and the American Academy of Pediatrics advocate for reducing pain in infants during procedures, recommending non-pharmacological methods as the first line of management. These methods, aimed at providing analgesic effects by creating a relaxing environment, are important because they do not have side effects. Some proven non-pharmacological techniques include breastfeeding, skin-to-skin contact, swaddling, music therapy, oral glucose, and pacifier use.

Music therapy is a widely used non-pharmacological method that helps reduce pain perception in newborns. Studies have shown its effectiveness in various settings. For instance, research with premature newborns found that music therapy during central venous catheter placement reduced physiological and behavioral reactions. Another study with 120 healthy newborns reported that having a musical baby crib mobile in vaccination rooms decreased pain levels and crying times. Other studies have similarly highlighted the positive effects of listening to or singing lullabies during painful procedures.

ELIGIBILITY:
Inclusion Criteria:

* born between 38-42 weeks,
* being 0-28 days,
* absence of visual and auditory problems,
* not using any pain reliever or sedative medication in the last four hours,
* parents' willingness to participate in the study,
* parents' knowledge of Turkish,
* parents' ability to read and write.

Exclusion Criteria:

* having a preterm birth,
* having a disease that causes chronic pain,
* having visual or auditory problems,
* using any pain or sedative medication in the last four hours.

Max Age: 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
ALPS-Neo pain and stress assessment scale | immediately after the intervention
  In this study, researchers used a mobile crib to help reduce pain in infants during needle procedures. Our primary outcome was the level of pain experienced by the infants. Pain was assessed using standardized pain assessment tools that are suitable for neonates. By comparing pain scores during the needle procedures, researchers aimed to determine the effectiveness of the mobile crib in reducing the infants' pain levels.

CONTACTS AND LOCATIONS:
Overall Officials: Eyşan Savaş, PhD, Principal Investigator — Koç University
Locations (1):
- Koc University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No